CLINICAL TRIAL: NCT00313378
Title: Effects of Perioperative Systemic Ketamine on Development of Long-term Neuropathic Pain After Thoracotomy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU63-0004
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Partial Pneumonectomy Under Lateral or Posterolateral Thoracotomy.
Keywords: Thoracotomy; Neuropathic pain; Nerve trauma; Ketamine; NMDA receptors
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- ketamine (Experimental): This study compares two groups of patients undergoing thoracotomy for partial pneumonectomy, one receiving intravenous ketamine since the beginning of procedure and then during 48 hours, the other receiving inactive normal saline (placebo).
  Interventions: Drug: Hypothetica
- placebo (Other): This study compares two groups of patients undergoing thoracotomy for partial pneumonectomy, one receiving intravenous ketamine since the beginning of procedure and then during 48 hours, the other receiving inactive normal saline (placebo).
  Interventions: Drug: Hypothetica

INTERVENTIONS:
Drug: Hypothetica

SUMMARY:
Lung surgery under thoracotomy is known to induce long-term pain which can be considered as neuropathic in many patients concerned [1,2]. The suspected origin of neuropathy is a direct traumatism of intercostal nerve(s) [3]. Among the possible preventive treatments that can be administered during the initial aggression, ketamine [4,5] appears as the easiest to use, as it is already commonly administered intra and postoperatively for improvement of analgesia [6].

DETAILED DESCRIPTION:
Lung surgery under thoracotomy is known to induce long-term pain which can be considered as neuropathic in many patients concerned [1,2]. The suspected origin of neuropathy is a direct traumatism of intercostal nerve(s) [3]. Among the possible preventive treatments that can be administered during the initial aggression, ketamine [4,5] appears as the easiest to use, as it is already commonly administered intra and postoperatively for improvement of analgesia [6]. This study compares two groups of patients undergoing thoracotomy for partial pneumonectomy, one receiving intravenous ketamine since the beginning of procedure and then during 48 hours, the other receiving inactive normal saline (placebo). The study is prospective, randomized, and double-blinded. The primary endpoint is to reduce chronic pain (on visual analogue scale) at the 4th month after surgery with ketamine. The objective is to obtain a mean value under 20/100 in the ketamine group, considering that the expected mean value for the control group is 38/100 (based on personal observations). The secondary endpoints are lower scores of neuropathic pain in the ketamine group, assessed by the NPSI questionnaire [7]. The impact of treatment on quality of life, assessed by a questionnaire (SF-36), is also studied. The data collected by clinical and psychophysical examination performed on all patients at the 4th month after surgery will be also considered for analysis, in order to understand better the features of post-thoracotomy neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* elective partial pneumonectomy under lateral or posterolateral thoracotomy, performed under standardized general anesthesia.

Exclusion Criteria:

* Patient's refusal
* Bad health status
* Previous neuropathic pain or treatment acting on neuropathic pain
* Major postoperative complication
* Intolerance to ketamine
* Epidural anesthesia

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2004-04; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Reduction of chronic pain

SECONDARY OUTCOMES:
Reduction of signs of neuropathic pain.
Improvement of quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Duale, Doctor, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Clermont-Ferrand University Hospital, Clermont-Ferrand, Auvergne, France

REFERENCES:
- [Background] Perttunen K, Tasmuth T, Kalso E. Chronic pain after thoracic surgery: a follow-up study. Acta Anaesthesiol Scand. 1999 May;43(5):563-7. doi: 10.1034/j.1399-6576.1999.430513.x. PMID 10342006
- [Background] Gotoda Y, Kambara N, Sakai T, Kishi Y, Kodama K, Koyama T. The morbidity, time course and predictive factors for persistent post-thoracotomy pain. Eur J Pain. 2001;5(1):89-96. doi: 10.1053/eujp.2001.0225. PMID 11394926
- [Background] Rogers ML, Henderson L, Mahajan RP, Duffy JP. Preliminary findings in the neurophysiological assessment of intercostal nerve injury during thoracotomy. Eur J Cardiothorac Surg. 2002 Feb;21(2):298-301. doi: 10.1016/s1010-7940(01)01104-6. PMID 11825739
- [Background] Felsby S, Nielsen J, Arendt-Nielsen L, Jensen TS. NMDA receptor blockade in chronic neuropathic pain: a comparison of ketamine and magnesium chloride. Pain. 1996 Feb;64(2):283-291. doi: 10.1016/0304-3959(95)00113-1. PMID 8740606
- [Background] Burton AW, Lee DH, Saab C, Chung JM. Preemptive intrathecal ketamine injection produces a long-lasting decrease in neuropathic pain behaviors in a rat model. Reg Anesth Pain Med. 1999 May-Jun;24(3):208-13. doi: 10.1016/s1098-7339(99)90129-3. PMID 10338169
- [Background] De Kock M, Lavand'homme P, Waterloos H. 'Balanced analgesia' in the perioperative period: is there a place for ketamine? Pain. 2001 Jun;92(3):373-380. doi: 10.1016/S0304-3959(01)00278-0. PMID 11376910
- [Background] Bouhassira D, Attal N, Fermanian J, Alchaar H, Gautron M, Masquelier E, Rostaing S, Lanteri-Minet M, Collin E, Grisart J, Boureau F. Development and validation of the Neuropathic Pain Symptom Inventory. Pain. 2004 Apr;108(3):248-257. doi: 10.1016/j.pain.2003.12.024. PMID 15030944
- [Result] Duale C, Sibaud F, Guastella V, Vallet L, Gimbert YA, Taheri H, Filaire M, Schoeffler P, Dubray C. Perioperative ketamine does not prevent chronic pain after thoracotomy. Eur J Pain. 2009 May;13(5):497-505. doi: 10.1016/j.ejpain.2008.06.013. Epub 2008 Sep 9. PMID 18783971
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/18783971